CLINICAL TRIAL: NCT06574620
Title: Accelerating the Actionability of Treatment in Resected and Locally Advanced Pancreatic Cancer
Brief Title: Using Tumour DNA and Proteins to Better Understand How Pancreatic Cancer Responds to Treatment
Acronym: ACCELERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Terry Fox Research Institute (Other); BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H24-01809
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Resectable Pancreatic Ductal Adenocarcinoma; Borderline Resectable Pancreatic Ductal Adenocarcinoma; Locally Advanced Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Genetic Testing; Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resectable Cohort (Other): Participants with resectable PDAC. Participants will provide tumour, fluid, and blood samples for genetic testing and other analyses. Tumour samples will be collected from standard resection surgery and optional biopsies. Fluid samples will be collected from a standard laparoscopy procedure. Blood samples will be collected at several timepoints throughout the study. Participants will receive standard chemotherapy (folinic acid (leucovorin), fluorouracil, irinotecan, and oxaliplatin (FOLFIRINOX) or gemcitabine-based) regimens.
  Interventions: Genetic: Genetic testing; Procedure: Optional biopsy; Procedure: Tissue collection
- Borderline Resectable Cohort (Other): Participants with borderline resectable PDAC. Participants will provide tumour, fluid, and blood samples for genetic testing and other analyses. Tumour samples will be collected from standard resection surgery and optional biopsies. Fluid samples will be collected from a standard laparoscopy procedure. Blood samples will be collected at several timepoints throughout the study. Participants will receive standard chemotherapy (FOLFIRINOX or gemcitabine-based) regimens.
  Interventions: Genetic: Genetic testing; Procedure: Optional biopsy; Procedure: Tissue collection
- Locally Advanced Cohort (Other): Participants with locally advanced PDAC. Participants will provide fluid and blood samples for genetic testing and other analyses. Fluid samples will be collected from a standard laparoscopy procedure. Blood samples will be collected at several timepoints throughout the study. Tumour samples may also be collected, if participants agree to optional biopsies. Participants will receive standard chemotherapy (FOLFIRINOX or gemcitabine-based) regimens.
  Interventions: Genetic: Genetic testing; Procedure: Optional biopsy; Procedure: Tissue collection

INTERVENTIONS:
Genetic: Genetic testing — Analyses of the deoxyribonucleic acid (DNA), ribonucleic acid (RNA), proteins, and other molecules in the sample.
Procedure: Optional biopsy — Optional collection of tumour tissue and normal tissue after the last dose of treatment.
Procedure: Tissue collection — Collection of tumour tissue and normal tissue from biopsy or standard resection surgery prior to the first dose of treatment.

SUMMARY:
The goal of this study is to learn if the genetic information and proteins from tumours can help treat pancreatic ductal adenocarcinoma (PDAC). The main questions it aims to answer are:

* Is it feasible to obtain genetic test results within a timeframe that can help inform treatment decisions for individuals with PDAC?
* Can the genetic test results provide information about how a tumour will respond to or resist treatment?

Participants will:

* Receive standard chemotherapy to treat their cancer.
* Provide samples of their blood, tissue, and fluid for genetic testing.
* Visit the clinic every 4 weeks for check-ups and tests.
* Complete questionnaires every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria prior to Pre-Baseline registration:

1. Age 18 years or older.
2. Histological or radiological diagnosis of resectable, borderline resectable, or locally advanced PDAC.
3. Medically fit and planned to undergo laparoscopic procedure as part of standard of care.
4. Able to give informed consent for the study-related procedures performed during laparoscopy.

Participants must meet all of the following criteria to be eligible for enrollment in the Main Study:

1. Age 18 years or older.
2. Enrolled in the Personalized Oncogenomics (POG) Program at BC Cancer.
3. Histological and/or radiological diagnosis of resectable, borderline resectable, or locally advanced PDAC. Participants without a histological diagnosis of PDAC must undergo confirmatory histological diagnosis prior to treatment start date.
4. Medically fit to undergo surgical resection of the primary lesion(s) as judged by the investigator (Resectable and Borderline Resectable Cohorts only).
5. Planned for adjuvant (Resectable and Borderline Resectable Cohorts) or first-line (Locally Advanced Cohort) therapy with FOLFIRINOX or a gemcitabine-based regimen, either as part of routine care or in combination with an investigational agent(s) within another clinical trial. Participants may have received pre-operative therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
7. Adequate organ function as defined by the following laboratory results obtained within 28 days prior to enrollment date:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L.
   2. Hemoglobin ≥ 9 g/dL.
   3. Platelets ≥ 75 x 10^9/L.
   4. Prothrombin time test and international normalized ratio (PT/INR) and partial thromboplastin time (PTT) ≤ 1.5 x Upper Limit of Normal (ULN).
   5. Total bilirubin ≤ 1.5 x ULN. Isolated bilirubin > 1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%.
   6. Aspartate aminotransferase (AST) and alanine aminotransferase (AST) ≤ 1.5 x ULN. If liver metastases are present, AST and ALT ≤ 5 x ULN is permitted.
   7. Albumin ≥ 25 g/L.
   8. One of the following:

      * Creatinine ≤ 1.5 x ULN.
      * Calculated creatinine clearance (as calculated by Cockcroft-Gault formula) ≥ 40 mL/min.
      * 24-hour urine creatinine clearance ≥ 40 mL/min.
8. Life expectancy greater than 90 days as judged by the investigator.
9. Able to give informed consent for the study procedures defined in this protocol.
10. Measurable disease by RECIST 1.1. For those in the Resectable and Borderline Resectable Cohorts, measurable disease must be present prior to resection surgery.

Exclusion Criteria:

1. Presence of distant or lymph node metastases. Individuals with metastatic PDAC are not eligible.
2. Currently receiving adjuvant (Resectable and Borderline Resectable Cohorts) or systemic (Locally Advanced Cohort) anti-cancer therapy (chemotherapy or any other anti-cancer agent) with one exception: pre-operative therapy is permitted.
3. Not fit for chemotherapy as judged by the investigator.
4. Presence of brain metastases.
5. Positive pregnancy test.
6. Unable to comply with the study assessments and procedures defined in this protocol.
7. Individuals who are otherwise judged by the investigator to be unfit to proceed with this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-28 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of comprehensive genomic results returned within 8 weeks of sample collection. | From the date of resection surgery or baseline ctDNA collection until genomic results are available (typically 8 weeks).
  The percentage of participants with comprehensive genomic results for their baseline tumour tissue and/or circulating tumour deoxyribonucleic acid (ctDNA) within 8 weeks of their collection.

SECONDARY OUTCOMES:
Overall response rate (ORR) in each study arm, as defined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 | From the date of the baseline scan (within 28 days of first dose) until the date of confirmed progression, withdrawal, date of death, or end of study, whichever comes first, assessed up to 72 months.
  The proportion of participants in each study arm who have a complete response (CR) or partial response (PR) to treatment, as defined by RECIST 1.1.
Disease control rate in each study arm, as defined by RECIST 1.1 | From the date of the baseline scan (within 28 days of first dose) until the date of confirmed progression, withdrawal, date of death, or end of study, whichever comes first, assessed up to 72 months.
  The proportion of participants in each study arm who have a complete response (CR), partial response (PR), or stable disease (SD) to treatment, as defined by RECIST 1.1.
Duration of response (DoR) in each study arm, as defined by RECIST 1.1 | From the first date of CR or PR until the first date of confirmed progression, withdrawal, date of death, or end of study, whichever comes first, assessed up to 72 months.
  The number of days between the first date of complete response (CR) or partial response (PR) and the earliest date of disease recurrence/progression or death due to any cause.
Progression-free survival (PFS) in each study arm from the initiation of chemotherapy | From the date of first dose of chemotherapy until the date of confirmed progression, withdrawal, date of death, or end of study, whichever comes first, assessed up to 72 months.
  The number of days from the first dose of chemotherapy until the date of progressive disease (PD), as defined by RECIST 1.1, for participants in each study arm.
Overall survival (OS) in each study arm from the initiation of chemotherapy | From the date of first dose of chemotherapy until the date of death or end of study, whichever comes first, assessed up to 72 months.]
  The number of days from the initiation of chemotherapy that participants survive in each study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Renouf, MD, Principal Investigator — BC Cancer
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Strickler JH, Satake H, George TJ, Yaeger R, Hollebecque A, Garrido-Laguna I, Schuler M, Burns TF, Coveler AL, Falchook GS, Vincent M, Sunakawa Y, Dahan L, Bajor D, Rha SY, Lemech C, Juric D, Rehn M, Ngarmchamnanrith G, Jafarinasabian P, Tran Q, Hong DS. Sotorasib in KRAS p.G12C-Mutated Advanced Pancreatic Cancer. N Engl J Med. 2023 Jan 5;388(1):33-43. doi: 10.1056/NEJMoa2208470. Epub 2022 Dec 21. PMID 36546651
- [Background] Wong HL, Zhao EY, Jones MR, Reisle CR, Eirew P, Pleasance E, Grande BM, Karasinska JM, Kalloger SE, Lim HJ, Shen Y, Yip S, Morin RD, Laskin J, Marra MA, Jones SJM, Schrader KA, Schaeffer DF, Renouf DJ. Temporal Dynamics of Genomic Alterations in a BRCA1 Germline-Mutated Pancreatic Cancer With Low Genomic Instability Burden but Exceptional Response to Fluorouracil, Oxaliplatin, Leucovorin, and Irinotecan. JCO Precis Oncol. 2018 Oct 19;2:PO.18.00057. doi: 10.1200/PO.18.00057. eCollection 2018. No abstract available. PMID 32913994
- [Background] O'Kane GM, Grunwald BT, Jang GH, Masoomian M, Picardo S, Grant RC, Denroche RE, Zhang A, Wang Y, Lam B, Krzyzanowski PM, Lungu IM, Bartlett JMS, Peralta M, Vyas F, Khokha R, Biagi J, Chadwick D, Ramotar S, Hutchinson S, Dodd A, Wilson JM, Notta F, Zogopoulos G, Gallinger S, Knox JJ, Fischer SE. GATA6 Expression Distinguishes Classical and Basal-like Subtypes in Advanced Pancreatic Cancer. Clin Cancer Res. 2020 Sep 15;26(18):4901-4910. doi: 10.1158/1078-0432.CCR-19-3724. Epub 2020 Mar 10. PMID 32156747
- [Background] Aung KL, Fischer SE, Denroche RE, Jang GH, Dodd A, Creighton S, Southwood B, Liang SB, Chadwick D, Zhang A, O'Kane GM, Albaba H, Moura S, Grant RC, Miller JK, Mbabaali F, Pasternack D, Lungu IM, Bartlett JMS, Ghai S, Lemire M, Holter S, Connor AA, Moffitt RA, Yeh JJ, Timms L, Krzyzanowski PM, Dhani N, Hedley D, Notta F, Wilson JM, Moore MJ, Gallinger S, Knox JJ. Genomics-Driven Precision Medicine for Advanced Pancreatic Cancer: Early Results from the COMPASS Trial. Clin Cancer Res. 2018 Mar 15;24(6):1344-1354. doi: 10.1158/1078-0432.CCR-17-2994. Epub 2017 Dec 29. PMID 29288237
- [Background] Neoptolemos JP, Palmer DH, Ghaneh P, Psarelli EE, Valle JW, Halloran CM, Faluyi O, O'Reilly DA, Cunningham D, Wadsley J, Darby S, Meyer T, Gillmore R, Anthoney A, Lind P, Glimelius B, Falk S, Izbicki JR, Middleton GW, Cummins S, Ross PJ, Wasan H, McDonald A, Crosby T, Ma YT, Patel K, Sherriff D, Soomal R, Borg D, Sothi S, Hammel P, Hackert T, Jackson R, Buchler MW; European Study Group for Pancreatic Cancer. Comparison of adjuvant gemcitabine and capecitabine with gemcitabine monotherapy in patients with resected pancreatic cancer (ESPAC-4): a multicentre, open-label, randomised, phase 3 trial. Lancet. 2017 Mar 11;389(10073):1011-1024. doi: 10.1016/S0140-6736(16)32409-6. Epub 2017 Jan 25. PMID 28129987
- [Background] Garcea G, Dennison AR, Pattenden CJ, Neal CP, Sutton CD, Berry DP. Survival following curative resection for pancreatic ductal adenocarcinoma. A systematic review of the literature. JOP. 2008 Mar 8;9(2):99-132. PMID 18326920
- [Background] Brenner DR, Poirier A, Woods RR, Ellison LF, Billette JM, Demers AA, Zhang SX, Yao C, Finley C, Fitzgerald N, Saint-Jacques N, Shack L, Turner D, Holmes E; Canadian Cancer Statistics Advisory Committee. Projected estimates of cancer in Canada in 2022. CMAJ. 2022 May 2;194(17):E601-E607. doi: 10.1503/cmaj.212097. PMID 35500919
- [Background] Jones MR, Williamson LM, Topham JT, Lee MKC, Goytain A, Ho J, Denroche RE, Jang G, Pleasance E, Shen Y, Karasinska JM, McGhie JP, Gill S, Lim HJ, Moore MJ, Wong HL, Ng T, Yip S, Zhang W, Sadeghi S, Reisle C, Mungall AJ, Mungall KL, Moore RA, Ma Y, Knox JJ, Gallinger S, Laskin J, Marra MA, Schaeffer DF, Jones SJM, Renouf DJ. NRG1 Gene Fusions Are Recurrent, Clinically Actionable Gene Rearrangements in KRAS Wild-Type Pancreatic Ductal Adenocarcinoma. Clin Cancer Res. 2019 Aug 1;25(15):4674-4681. doi: 10.1158/1078-0432.CCR-19-0191. Epub 2019 May 8. PMID 31068372
- [Background] Aguirre AJ. Oncogenic NRG1 Fusions: A New Hope for Targeted Therapy in Pancreatic Cancer. Clin Cancer Res. 2019 Aug 1;25(15):4589-4591. doi: 10.1158/1078-0432.CCR-19-1280. Epub 2019 Jun 4. PMID 31164372
- [Background] Oettle H, Neuhaus P, Hochhaus A, Hartmann JT, Gellert K, Ridwelski K, Niedergethmann M, Zulke C, Fahlke J, Arning MB, Sinn M, Hinke A, Riess H. Adjuvant chemotherapy with gemcitabine and long-term outcomes among patients with resected pancreatic cancer: the CONKO-001 randomized trial. JAMA. 2013 Oct 9;310(14):1473-81. doi: 10.1001/jama.2013.279201. PMID 24104372
- [Background] Ferrone CR, Pieretti-Vanmarcke R, Bloom JP, Zheng H, Szymonifka J, Wargo JA, Thayer SP, Lauwers GY, Deshpande V, Mino-Kenudson M, Fernandez-del Castillo C, Lillemoe KD, Warshaw AL. Pancreatic ductal adenocarcinoma: long-term survival does not equal cure. Surgery. 2012 Sep;152(3 Suppl 1):S43-9. doi: 10.1016/j.surg.2012.05.020. Epub 2012 Jul 3. PMID 22763261
- [Background] Goldstein D, El-Maraghi RH, Hammel P, Heinemann V, Kunzmann V, Sastre J, Scheithauer W, Siena S, Tabernero J, Teixeira L, Tortora G, Van Laethem JL, Young R, Penenberg DN, Lu B, Romano A, Von Hoff DD. nab-Paclitaxel plus gemcitabine for metastatic pancreatic cancer: long-term survival from a phase III trial. J Natl Cancer Inst. 2015 Jan 31;107(2):dju413. doi: 10.1093/jnci/dju413. Print 2015 Feb. PMID 25638248
- [Background] Canadian Cancer Society's Advisory Committee on Cancer Statistics. Canadian Cancer Statistics 2017: 1-142. Toronto, ON: Canadian Cancer Society; 2017.
- [Background] Conroy T, Desseigne F, Ychou M, Bouche O, Guimbaud R, Becouarn Y, Adenis A, Raoul JL, Gourgou-Bourgade S, de la Fouchardiere C, Bennouna J, Bachet JB, Khemissa-Akouz F, Pere-Verge D, Delbaldo C, Assenat E, Chauffert B, Michel P, Montoto-Grillot C, Ducreux M; Groupe Tumeurs Digestives of Unicancer; PRODIGE Intergroup. FOLFIRINOX versus gemcitabine for metastatic pancreatic cancer. N Engl J Med. 2011 May 12;364(19):1817-25. doi: 10.1056/NEJMoa1011923. PMID 21561347
- [Background] Conroy T, Hammel P, Hebbar M, Ben Abdelghani M, Wei AC, Raoul JL, Chone L, Francois E, Artru P, Biagi JJ, Lecomte T, Assenat E, Faroux R, Ychou M, Volet J, Sauvanet A, Breysacher G, Di Fiore F, Cripps C, Kavan P, Texereau P, Bouhier-Leporrier K, Khemissa-Akouz F, Legoux JL, Juzyna B, Gourgou S, O'Callaghan CJ, Jouffroy-Zeller C, Rat P, Malka D, Castan F, Bachet JB; Canadian Cancer Trials Group and the Unicancer-GI-PRODIGE Group. FOLFIRINOX or Gemcitabine as Adjuvant Therapy for Pancreatic Cancer. N Engl J Med. 2018 Dec 20;379(25):2395-2406. doi: 10.1056/NEJMoa1809775. PMID 30575490
- [Background] Moore MJ, Goldstein D, Hamm J, Figer A, Hecht JR, Gallinger S, Au HJ, Murawa P, Walde D, Wolff RA, Campos D, Lim R, Ding K, Clark G, Voskoglou-Nomikos T, Ptasynski M, Parulekar W; National Cancer Institute of Canada Clinical Trials Group. Erlotinib plus gemcitabine compared with gemcitabine alone in patients with advanced pancreatic cancer: a phase III trial of the National Cancer Institute of Canada Clinical Trials Group. J Clin Oncol. 2007 May 20;25(15):1960-6. doi: 10.1200/JCO.2006.07.9525. Epub 2007 Apr 23. PMID 17452677
- [Background] Seicean A, Petrusel L, Seicean R. New targeted therapies in pancreatic cancer. World J Gastroenterol. 2015 May 28;21(20):6127-45. doi: 10.3748/wjg.v21.i20.6127. PMID 26034349
- [Background] Collisson EA, Bailey P, Chang DK, Biankin AV. Molecular subtypes of pancreatic cancer. Nat Rev Gastroenterol Hepatol. 2019 Apr;16(4):207-220. doi: 10.1038/s41575-019-0109-y. PMID 30718832
- [Background] Waddell N, Pajic M, Patch AM, Chang DK, Kassahn KS, Bailey P, Johns AL, Miller D, Nones K, Quek K, Quinn MC, Robertson AJ, Fadlullah MZ, Bruxner TJ, Christ AN, Harliwong I, Idrisoglu S, Manning S, Nourse C, Nourbakhsh E, Wani S, Wilson PJ, Markham E, Cloonan N, Anderson MJ, Fink JL, Holmes O, Kazakoff SH, Leonard C, Newell F, Poudel B, Song S, Taylor D, Waddell N, Wood S, Xu Q, Wu J, Pinese M, Cowley MJ, Lee HC, Jones MD, Nagrial AM, Humphris J, Chantrill LA, Chin V, Steinmann AM, Mawson A, Humphrey ES, Colvin EK, Chou A, Scarlett CJ, Pinho AV, Giry-Laterriere M, Rooman I, Samra JS, Kench JG, Pettitt JA, Merrett ND, Toon C, Epari K, Nguyen NQ, Barbour A, Zeps N, Jamieson NB, Graham JS, Niclou SP, Bjerkvig R, Grutzmann R, Aust D, Hruban RH, Maitra A, Iacobuzio-Donahue CA, Wolfgang CL, Morgan RA, Lawlor RT, Corbo V, Bassi C, Falconi M, Zamboni G, Tortora G, Tempero MA; Australian Pancreatic Cancer Genome Initiative; Gill AJ, Eshleman JR, Pilarsky C, Scarpa A, Musgrove EA, Pearson JV, Biankin AV, Grimmond SM. Whole genomes redefine the mutational landscape of pancreatic cancer. Nature. 2015 Feb 26;518(7540):495-501. doi: 10.1038/nature14169. PMID 25719666
- [Background] O'Reilly EM, Lee JW, Zalupski M, Capanu M, Park J, Golan T, Tahover E, Lowery MA, Chou JF, Sahai V, Brenner R, Kindler HL, Yu KH, Zervoudakis A, Vemuri S, Stadler ZK, Do RKG, Dhani N, Chen AP, Kelsen DP. Randomized, Multicenter, Phase II Trial of Gemcitabine and Cisplatin With or Without Veliparib in Patients With Pancreas Adenocarcinoma and a Germline BRCA/PALB2 Mutation. J Clin Oncol. 2020 May 1;38(13):1378-1388. doi: 10.1200/JCO.19.02931. Epub 2020 Jan 24. PMID 31976786
- [Background] Sener SF, Fremgen A, Menck HR, Winchester DP. Pancreatic cancer: a report of treatment and survival trends for 100,313 patients diagnosed from 1985-1995, using the National Cancer Database. J Am Coll Surg. 1999 Jul;189(1):1-7. doi: 10.1016/s1072-7515(99)00075-7. PMID 10401733
- [Background] Oettle H, Post S, Neuhaus P, Gellert K, Langrehr J, Ridwelski K, Schramm H, Fahlke J, Zuelke C, Burkart C, Gutberlet K, Kettner E, Schmalenberg H, Weigang-Koehler K, Bechstein WO, Niedergethmann M, Schmidt-Wolf I, Roll L, Doerken B, Riess H. Adjuvant chemotherapy with gemcitabine vs observation in patients undergoing curative-intent resection of pancreatic cancer: a randomized controlled trial. JAMA. 2007 Jan 17;297(3):267-77. doi: 10.1001/jama.297.3.267. PMID 17227978
- [Background] Chan-Seng-Yue M, Kim JC, Wilson GW, Ng K, Figueroa EF, O'Kane GM, Connor AA, Denroche RE, Grant RC, McLeod J, Wilson JM, Jang GH, Zhang A, Dodd A, Liang SB, Borgida A, Chadwick D, Kalimuthu S, Lungu I, Bartlett JMS, Krzyzanowski PM, Sandhu V, Tiriac H, Froeling FEM, Karasinska JM, Topham JT, Renouf DJ, Schaeffer DF, Jones SJM, Marra MA, Laskin J, Chetty R, Stein LD, Zogopoulos G, Haibe-Kains B, Campbell PJ, Tuveson DA, Knox JJ, Fischer SE, Gallinger S, Notta F. Transcription phenotypes of pancreatic cancer are driven by genomic events during tumor evolution. Nat Genet. 2020 Feb;52(2):231-240. doi: 10.1038/s41588-019-0566-9. Epub 2020 Jan 13. PMID 31932696
- [Background] Karasinska JM, Topham JT, Kalloger SE, Jang GH, Denroche RE, Culibrk L, Williamson LM, Wong HL, Lee MKC, O'Kane GM, Moore RA, Mungall AJ, Moore MJ, Warren C, Metcalfe A, Notta F, Knox JJ, Gallinger S, Laskin J, Marra MA, Jones SJM, Renouf DJ, Schaeffer DF. Altered Gene Expression along the Glycolysis-Cholesterol Synthesis Axis Is Associated with Outcome in Pancreatic Cancer. Clin Cancer Res. 2020 Jan 1;26(1):135-146. doi: 10.1158/1078-0432.CCR-19-1543. Epub 2019 Sep 3. PMID 31481506
- [Background] Golan T, Hammel P, Reni M, Van Cutsem E, Macarulla T, Hall MJ, Park JO, Hochhauser D, Arnold D, Oh DY, Reinacher-Schick A, Tortora G, Algul H, O'Reilly EM, McGuinness D, Cui KY, Schlienger K, Locker GY, Kindler HL. Maintenance Olaparib for Germline BRCA-Mutated Metastatic Pancreatic Cancer. N Engl J Med. 2019 Jul 25;381(4):317-327. doi: 10.1056/NEJMoa1903387. Epub 2019 Jun 2. PMID 31157963